CLINICAL TRIAL: NCT05942690
Title: Ultrasound Evaluation of Diaphragmatic Contractility After Manual Osteopathic Intervention in Professional Handball Players: a Pilot Study
Brief Title: Osteopathic Intervention in Professional Handball Players
Acronym: ECHODIAPOST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no more possibly to include subjects (subject unavailability)
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/23/0146
Record Dates: First submitted 2023-06-23; First posted 2023-07-12 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Osteopathia
Keywords: diaphragm; ultrasound; contractibility; osteopathic intervention
MeSH Terms: conditions — Bone Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental (Experimental): The intervention evaluated is a technique of prolonged abdominal manual pressure centered on the zone of restriction of mobility called "trigger point" with diaphragmatic aim.
  Interventions: Procedure: manual osteopathic intervention

INTERVENTIONS:
Procedure: manual osteopathic intervention — The subject sits on the examination table for the manual osteopathic intervention. The expert osteopath, having no report from the sonographers, will manually test breathing diaphragmatic and will bring osteopathic manual treatment to the area of mobility restriction

SUMMARY:
The aim is to study the effectiveness of a common osteopathic intervention in professional handball players on diaphragmatic contractility and its correlations with posture. This study has never been done in healthy subjects. It is a scientific process of objectification of an osteopathic technique commonly performed in this population. The main objective is to assess diaphragmatic contractibility using ultrasound after abdominal osteopathic intervention (OMT).

DETAILED DESCRIPTION:
The context is that of optimizing the performance of professional handball players. The aim is to study the effectiveness of a common osteopathic intervention in professional handball players on diaphragmatic contractility and its correlations with posture. This study has never been done in healthy subjects. It is a scientific process of objectification of an osteopathic technique commonly performed in this population.

The main objective is to assess diaphragmatic contractibility after abdominal osteopathic intervention (OMT).

The secondary objective is to evaluate the impact of this manual intervention in professional handball players on:

* other diaphragmatic ultrasound data
* on spirometry
* postural control

Prospective pilot non-interventional controlled monocentric study opened in healthy male and female International players who are part of the French Handball team. Approach to objectification of current practice.

ELIGIBILITY:
Inclusion Criteria:

* healthy male and female International players who are part of the French Handball team

Exclusion Criteria:

* history of thoracic or diaphragmatic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-07-30 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Variation in the fraction of diaphragm thickening (right and left) measured on ultrasound before and after the procedure | Day 1
  The subject undergoes the ultrasound which will investigate the contractility of the diaphragm muscle. Two expert sonographers from G-ECHO will perform the ultrasound on each of the athletes, and note 3 successive measurements to check the stability of the results.

SECONDARY OUTCOMES:
expiratory diaphragmatic thickness | Day 1
  expiratory diaphragmatic thickness will be measured by echography (mm) after manual abdominal osteopathic intervention
Variation of the Forced Vital Capacity (FVC) measured in spirometry before and after the intervention | Day 1
  The subject performs spirometry while standing with a Spirobank spirometer. 3 successive measurements keeping only the highest value.
Postural analysis | Day 2
  postural analysis will be perform using Cyber-Sabot type platform. the measurements will be done at day 1 before manual abdominal osteopathic intervention and at day 2
Inspiratory diaphragmatic thickness | day 1
  Inspiratory diaphragmatic thickness will be measured by echography (mm) after manual abdominal osteopathic intervention
diaphragmatic contraction velocity | day 1
  Diaphragmatic contraction velocity is expressed in % will be measured by echography after manual abdominal osteopathic intervention
diaphragmatic amplitude | day 1
  Diaphragmatic amplitude is expressed in mm and will be measured by echography after manual abdominal osteopathic intervention

CONTACTS AND LOCATIONS:
Overall Officials: Elise NOEL-SAVINA, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Maison du Handball, Créteil, France